CLINICAL TRIAL: NCT05379530
Title: Thromboelastography (TEG) and Intraoperative Coagulation Management of Pediatric Patients Undergoing Procedures With High Anticipated Blood Loss
Brief Title: TEG Use in Children Undergoing Procedures With High Anticipated Blood Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Goobie, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P00040518
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Surgical Blood Loss; Surgical Hemorrhage; Post Operative Hemorrhage
Keywords: thromboelastography; blood transfusion; viscoelastic test-guided; massive hemorrhage
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Thrombelastography

STUDY DESIGN:
Intervention Model Description: Thromboelastography (TEG) analysis will be done on all subjects who consent to participate in the study. TEG results will be made available to the anesthesiologist caring for the subject and may be used to help guide their care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEG Arm (Experimental): All patients enrolled in the study will have up to four 0.5cc blood samples obtained specifically for TEG analysis at the following defined points (for a total of up to 2cc of blood) when other routine labs are drawn (via an existing intravenous line or arterial line placed for clinical care) :
  * Once at the beginning of the case
  * Once at the end of the case
  * Up to two times at the same time as arterial blood gas (ABG) samples (if drawn)
  The research team will collect the following information from the electronic medical record and input it into the Internal REDCap database:
  * De-identified demographic data, including age, height, weight, and diagnosis
  * Preoperative, intraoperative, and postoperative laboratory values( including PT, PTT, INR and fibrinogen and platelets), as dictated by standard clinical practice
  * Time of TEG results printed and time delivered to anesthesiologist
  * Complications/Adverse events within the first 48 hours postoperatively
  Interventions: Diagnostic Test: Thromboelastography (TEG); Other: Anesthesia Provider Survey

INTERVENTIONS:
Diagnostic Test: Thromboelastography (TEG) — Thromboelastography (TEG) is a type of Viscoelastic testing (ROTEM is another example) and is a validated point of care method of dynamically assessing intraoperative coagulopathy via functional assay.
Other: Anesthesia Provider Survey — Pre-operative and post-operative provider surveys will be distributed to anesthesiologists caring for study subjects to assess knowledge, practice, and attitudes about TEG.

SUMMARY:
The research team proposes a prospective, observational study to better understand how TEG can be useful in guiding clinical practice in the Main OR for subject's undergoing high transfusion risk surgeries.

Intraoperatively, transfusion of blood products is frequently required to restore oxygen carrying capacity, perfusion and improve coagulation. Both under and over transfusion pose significant risks, particularly to pediatric patients with small starting intravascular volumes. Thromboelastography (TEG) is a validated method of dynamically assessing intraoperative coagulopathy via functional assay. However, while FDA approved and widely used in the adult setting, TEG is not commonly utilized in the setting of bleeding pediatric patients.

Recently, TEG has been made available at BCH for clinical purposes and is being used solely in the cardiac surgery setting. The investigators aim to provide TEG data for non-cardiac pediatric surgical cases with a high risk of intraoperative blood loss in order to assess the impact of this tool on intraoperative management.

DETAILED DESCRIPTION:
Intraoperatively, transfusion of blood products is frequently required to restore oxygen carrying capacity, perfusion and improve coagulation. Both under and over transfusion pose significant risks, particularly to pediatric patients with small starting intravascular volumes. Thromboelastography (TEG) is a type of Viscoelastic testing (ROTEM is another example) and is a validated point of care method of dynamically assessing intraoperative coagulopathy via functional assay. It provides more useful information than the commonly used laboratory values of INR, PT, PTT and Fibrinogen. However, while FDA approved and widely used in the adult setting, TEG is not commonly utilized in the setting of bleeding pediatric patients. Recently, TEG has been made available at Boston Children's Hospital (BCH) for clinical purposes exclusively in the cardiac surgery setting. The investigators aim to provide TEG data for general main operating room (MOR) pediatric surgical cases with a high risk of intraoperative blood loss in order to assess the impact of this tool on intraoperative management of the bleeding patient.

Primary Aim:

Assess the efficacy of providing real time viscoelastic testing (TEG) to anesthesiologists managing of pediatric patients with hemostatic bleeding undergoing procedures with high historical rates of blood transfusions. The outcome will be perioperative (intraoperative and within 24 H postoperative) hemostatic blood product transfusion (type of blood product and volume mL/g) within specific high blood loss surgical procedures. Data will be compared to matched cohorts using historical data from the same surgery types available in the Department of Anesthesia Blood Management Database.

Secondary Aim:

Assess the feasibility of providing real time and interpreting TEG data in a busy, academic, pediatric main OR at relevant clinical time points. Pre-operative and post-operative surveys will be administered to clinicians to gauge interest and knowledge in using TEG.

Hypothesis

The hypothesis is that the availability of TEG to help the management of pediatric surgical patients at a high risk for blood loss will improve targeted transfusion management, decrease overall intraoperative blood product utilization, and decrease variability in care. This data may ultimately yield future BCH viscoelastic test-guided (VET) transfusion protocols allowing a goal-directed approach. Benefits from this approach might translate into:

I. less exposure of the pediatric patient to blood products, thereby reducing the inherent risks of transfusion such as transfusion reactions, blood product associated infections and TRALI/TACO II. a reduction in costs, and III. Identification of clinical processes, such as fibrinolysis, that might otherwise be missed, leading to specific interventions (e.g. use of antifibrinolytics).

Although different blood product transfusion algorithms have been described in different clinical settings, there are no current VET (TEG or ROTEM) protocols in use for pediatric MOR surgical patients at this single center. See Appendix A for both existing BCH massive hemorrhage guidelines (MHG) and a massive hemorrhage protocol (MHP) including VET guided care - published as a supplement to the 2019 Society for the advancement of blood management administrative and clinical standards for patient blood management programs publication6.

These VET MHG will be available to the providers to help diagnosis and guide hemostatic blood product transfusion management intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing non-cardiac surgery at BCH with a high likelihood of blood transfusion. Specifically these are defined as a surgery with greater than 25% likelihood of transfusion of any non-albumin blood product.
* Eligible surgeries include:
* spinal surgery
* laparotomy
* liver transplant
* craniofacial surgery
* esophageal atresia
* craniotomy/hemispherectomy
* major abdominal surgery
* major hip surgery
* major plastic surgery

Exclusion Criteria:

* Patients undergoing cardiac surgery or ECMO cannulation, as these surgeries are generally considered outside the scope of general pediatric surgery.
* Patients presenting for emergent surgery
* Patients undergoing surgeries off hours (between 8pm and 8 am), when TEG analysis is unobtainable

Max Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of utilizing Viscoelastic testing (Thromboelastography;TEG) to diagnose and guide management as measured by type of hemostatic blood products transfused. | 1 year
  Assess the efficacy of utilizing Viscoelastic testing (TEG) in the diagnosis and management of hemostatic bleeding intraoperatively and compare to the current standard hemostatic product transfusion practice on the management of pediatric patients undergoing specific non-cardiac surgical procedures with high historical rates of transfusions at a single center. The efficacy of TEG will be measured in types of hemostatic blood products (fresh frozen plasma, platelets, cryoprecipitate) transfused within specific high blood loss surgical procedures as compared to historical matches controls which is available in the Department of Anesthesiology Patient Blood Management Database.
Efficacy of utilizing Viscoelastic testing (TEG) to diagnose and guide intraoperative management as measured by amount (mL/kg) hemostatic blood products transfused. | 1 year
  Assess the efficacy of utilizing Viscoelastic testing (TEG) in the diagnosis and management of hemostatic bleeding in specific surgical cohorts and compare to the current standard hemostatic product transfusion practice on the management of pediatric patients undergoing specific non-cardiac surgical procedures with high historical rates of transfusions at BCH. The efficacy of TEG will be measured in amount (mL/kg) of hemostatic blood products (fresh frozen plasma, platelets, cryoprecipitate) transfused within specific high blood loss surgical procedures as compared to historical transfusion data ( and standard laboratory data including PT, PTT, INR and fibrinogen and platelets) for the same surgery types available in the Department of Anesthesiology Patient Blood Management Database.

SECONDARY OUTCOMES:
Assess the feasibility of providing and interpreting TEG data in a busy, academic, pediatric non-cardiac operating room | 1 year
  Assess the feasibility of providing and interpreting TEG data in a busy, academic, pediatric non-cardiac operating room at relevant clinical time points. Pre-operative and post-operative provider surveys will be distributed to assess knowledge, practice, and attitudes. Surveys responses will be free-form and multiple choice.
Red blood cell transfusion amounts | 1 year
  The investigators will also compare red blood cell transfusion (mL/kg) amounts within the specific surgical cohorts between the TEG group and historical matched transfusion data.
Tranexamic acid (TXA) use | 1 year
  The investigators will compare tranexamic (TXA) use within specific cohorts between the TEG group and historical matched transfusion data.
Cell salvage use | 1 year
  The investigators will compare cell salvage use within specific cohorts between the TEG group and historical matched transfusion data.

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other researchers.